CLINICAL TRIAL: NCT00616798
Title: Randomized, Double-blind, Placebo-controlled add-on Trial of the Safety and Efficacy of RO4917838 in Outpatients on Select Atypical Antipsychotics With Prominent Negative or Disorganized Thought Symptoms
Brief Title: A Study of RO4917838 in Combination With Antipsychotic Treatment in Patients With Schizophrenia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN20372
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 3 (Experimental)
  Interventions: Drug: RO4917838; Drug: Standard antipsychotic therapy
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Standard antipsychotic therapy
- 1 (Experimental)
  Interventions: Drug: RO4917838; Drug: Standard antipsychotic therapy
- 2 (Experimental)
  Interventions: Drug: RO4917838; Drug: Standard antipsychotic therapy

INTERVENTIONS:
Drug: RO4917838 — 10mg po daily
  Arms: 1
Drug: RO4917838 — 30mg po daily
  Arms: 2
Drug: RO4917838 — 60mg po daily
  Arms: 3
Drug: Placebo — po daily
  Arms: 4
Drug: Standard antipsychotic therapy — As prescribed

SUMMARY:
This study will determine the efficacy and safety of RO4917838 in patients with schizophrenia who are stable on current antipsychotic treatment (olanzapine, que tiapine, risperidone, paliperidone or aripiprazole) with prominent negative or d isorganized thought symptoms. After a 4 week run in period on their current anti psychotic treatment, patients will be randomized to receive placebo 10mg, 30mg, or 60mg of RO4917838 once daily, p.o., as add-on therapy. The anticipated time o n study treatment is <3 months, and the target sample size is 100-500 individual s.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-60 years of age;
* diagnosis of schizophrenia (based on screening tests);
* outpatients, with no hospitalization for worsening of schizophrenia within 3 months;
* medically and psychiatrically stable over prior 1 month and psychiatrically stable without symptom exacerbation within prior 3 months;
* currently taking no more than 2 antipsychotic drugs.

Exclusion Criteria:

* began a new non-medication treatment for schizophrenia or other psychiatric condition within last 3 months;
* on >1 antidepressant, or a change in dose of antidepressant within 3 months;
* alcohol or substance abuse or dependence within 3 months;
* has previously received RO4917838.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in PANSS (Positive and Negative Syndrome Scale) negative factor score. | Week 8

SECONDARY OUTCOMES:
Change from baseline in total PANSS score, CGI, PSP, SGLS; cognition status changes. | Throughout study
AEs, laboratory parameters, C-SSRS | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- United States (13):
  - Granada Hills, California
  - Los Angeles, California
  - Oceanside, California
  - Torrance, California
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Brooklyn, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - DeSoto, Texas
  - Irving, Texas
- Vienna, Austria
- Brazil (5):
  - Curitiba
  - Pelotas
  - Rio de Janeiro
  - Salvador
  - São Paulo
- France (3):
  - Marseille
  - Orvault
  - Toulon
- Germany (6):
  - Achim
  - Bochum
  - Freiburg im Breisgau
  - Hamburg
  - Nuremberg
  - Westerstede
- Hungary (5):
  - Balassagyarmat
  - Budapest
  - GYR
  - Gyula
  - Nyíregyháza
- Japan (10):
  - Aichi
  - Chiba
  - Fukuoka
  - Gunma
  - Kanagawa
  - Nagasaki
  - Saga
  - Sapporo
  - Tokushima
  - Tokyo
- Mexico (2):
  - Mexico City
  - Monterrey
- Poland (6):
  - Bydgoszcz
  - Kielce
  - Skorzewo
  - Torun
  - Tuszyn
  - Żuromin
- Russia (5):
  - Kazan'
  - Lipetsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg

REFERENCES:
- [Derived] Umbricht D, Alberati D, Martin-Facklam M, Borroni E, Youssef EA, Ostland M, Wallace TL, Knoflach F, Dorflinger E, Wettstein JG, Bausch A, Garibaldi G, Santarelli L. Effect of bitopertin, a glycine reuptake inhibitor, on negative symptoms of schizophrenia: a randomized, double-blind, proof-of-concept study. JAMA Psychiatry. 2014 Jun;71(6):637-46. doi: 10.1001/jamapsychiatry.2014.163. PMID 24696094